CLINICAL TRIAL: NCT06768554
Title: Retrospective Analysis of Prognostic Indicators of Diabetic Foot Ulcer
Brief Title: Predictive Analysis of Diabetic Foot Ulcer
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Ruijin Hospital
Other Study IDs: CCEMD-20241001
Record Dates: First submitted 2024-12-10; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Diabetic Foot Disease; Diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Hemoglobin A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Level of blood sugar control (e.g., hemoglobin A1C), severity of infection, blood supply status, and other complications (e.g., peripheral neuropathy) — Level of blood sugar control (e.g., hemoglobin A1C), severity of infection, blood supply status, and other complications (e.g., peripheral neuropathy)

SUMMARY:
The purpose of this study was to retrospectively analyze the wound condition, limb condition, ulcer recurrence and cardiovascular and mortality of patients with diabetic foot ulcer after admission to our hospital from 2009 to 2014, so as to understand the changes in the condition of patients with diabetic foot ulcer after treatment, provide evidence for the treatment of diabetic foot, and clarify the risk of diagnosis and treatment of diabetic foot.

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) is one of the most common and serious complications in patients with diabetes. Due to its high incidence and complicated treatment process, DFU often has a significant impact on patients' quality of life. In order to gain an in-depth understanding of the wound changes of diabetic foot patients after admission, this study aims to systematically analyze the data of the database of diabetic foot patients in Ruijin Hospital, analyze the wound healing, ulcer recurrence and limb changes of diabetic foot patients, including amputation and other conditions, and then further determine the main factors affecting diabetic foot ulcer healing. Guide clinicians to develop more effective treatment plans; Provide data support to help optimize the treatment flow of diabetic foot and reduce length of stay and recurrence rates; To improve the overall treatment effect of diabetic foot patients and improve their quality of life.

Objective:

1. The wound condition, limb condition, ulcer recurrence and cardiovascular and mortality changes of patients with diabetic foot after treatment were analyzed to clarify the risk of diagnosis and treatment of the disease and provide evidence for the treatment of diabetic foot.
2. To assess the progress of wound healing in patients with diabetic foot after admission to hospital and identify key factors that promote or delay healing.
3. By comparing the effects of different treatment methods (such as drug therapy, surgical intervention, adjuvant therapy, etc.), the most suitable treatment strategy is found.
4. The incidence of complications during and after treatment was analyzed, and effective management strategies were discussed.

Methods:Through systematic analysis of the data from the database of diabetic foot patients in Ruijin Hospital, the wound healing, ulcer recurrence and limb changes of diabetic foot patients, including amputation, were analyzed, and then the main factors affecting diabetic foot ulcer healing were further determined.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Gender: males and females
3. Patients diagnosed with diabetic foot ulcers (including those on the Wagner scale 0-5)
4. Receive inpatient treatment during the designated study period

Exclusion Criteria:

1. Patients with severe systemic disease (such as end-stage renal disease, advanced cancer, etc.) may have influenced the study results
2. Patients unable to complete follow-up or with incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic foot ulcer patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer healing rate in diabetic foot ulcers | Look at the last 10 years retrospectively
Ulcer recurrence rate in diabetic foot ulcer patients | Look at the last 10 years retrospectively
Amputation rate in diabetic foot ulcers | Look at the last 10 years retrospectively
Mortality of diabetic foot ulcers | Look at the last 10 years retrospectively

SECONDARY OUTCOMES:
Key independent factors that affect wound healing | Look at the last 10 years retrospectively
  Through in-depth analysis of the diabetic foot ulcer patient database, the study is expected to identify key independent factors that affect wound healing, including the patient's level of blood sugar control (such as hemoglobin A1C), severity of infection, blood supply status, and other complications (such as peripheral neuropathy and vascular disease).

CONTACTS AND LOCATIONS:
Locations (1):
- National Clinical Medical Research Center for Metabolic Diseases (Shanghai), Shanghai, China